CLINICAL TRIAL: NCT03805724
Title: Is Entamoeba Gingivalis A Risk Factor In Periodontal Diseases
Brief Title: Entamoeba Gingivalis and Periodontal Disease
Status: Completed | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Gihane Gharib Madkour, Associate Professor, Cairo University
Other Study IDs: 15062006
Record Dates: First submitted 2019-01-11; First posted 2019-01-16 (Actual); Last update posted 2019-04-02 (Actual); Status verified 2019-03

CONDITIONS: Periodontal Diseases
MeSH Terms: conditions — Periodontal Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 2 Weeks
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Periodontally healthy subjects: They will be selected from healthy subjects who attend the restorative dental clinic and has clinically healthy gingiva with zero plaque index, gingival index and clinical attachment level & probing depth ≤ 3 mm. Plaque samples will be collected.
  Interventions: Other: Plaque Samples
- Chronic Periodontitis: Chronic periodontitis patients having probing depth of ≥3 mm and clinical attachment level ≥ 1 mm. Plaque samples will be collected.
  Interventions: Other: Plaque Samples
- Chronic Gingivitis: Gingivitis patients having signs of clinical inflammation with no clinical attachment loss. Plaque samples will be collected
  Interventions: Other: Plaque Samples

INTERVENTIONS:
Other: Plaque Samples — After carefully drying of the selected site and isolation by cotton roll, plaque samples will be collected by sweeping movement of the probe at gingival crevices of the tooth aspect with pervious inclusion criteria for obtaining of the plaque sample. Samples will be immediately dipped in sterile Eppendorf tubes containing PVA.

SUMMARY:
This current study aims to clarify the relationship between the occurrence of Entamoeba gingivalis infection and the specter of gingivitis & chronic periodontitis among Egyptian patients in comparison to healthy volunteers as a control group.

DETAILED DESCRIPTION:
Three groups will be included in the current study. 40 Plaque samples will be collected from gingivitis patients (group 1), 40 from chronic periodontitis patients (group 2) plus 40 samples from healthy volunteers (group 3). Diagnosis of parasitic stages will rely on direct microscopic detection using permanent stains, Trichrome stain and haematoxylin and eosin stain in addition to direct wet mount examination.

ELIGIBILITY:
Inclusion Criteria:

* Chronic Gingivitis patients with signs of clinical inflammation with no clinical attachment loss.
* Chronic Periodontitis patients having probing depth of ≥3 mm and clinical attachment level ≥ 1 mm.
* The control group: healthy subjects who attend the restorative dental clinic and had clinically healthy gingiva.

Exclusion Criteria:

* Patients with any systemic diseases

Ages: 35 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Gingivitis & Chronic periodontitis patients will be selected from the outpatients Clinic, Department of Oral Medicine, Periodontology and Diagnosis, Faculty of Dentistry, Fayoum University. Clinical examination for all patients will be performed including the following periodontal parameters: plaque index, gingival index, probing depth, and clinical attachment level. These measurements will be recorded by a single calibrated expert examiner at six sites for all teeth (mesiobuccal, mesiolingual, midbuccal, distobuccal, distolingual, and midlingual). PI is assessed by measuring the presence or absence of supragingival biofilm with a sweeping movement of the probe around the surfaces of all teeth
Sampling Method: Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2018-07-13 (Actual); Primary Completion 2019-01-18 (Actual); Study Completion 2019-01-18 (Actual)

PRIMARY OUTCOMES:
Presence of Entamoaba Gingivalis parasite in dental plaque assessed by direct microscopic examination | 2 weeks
  Direct microscopic detection of Entamoaba Gingivalis in dental plaque samples using Trichrome stain

CONTACTS AND LOCATIONS:
Overall Officials: Gihane G Madkour, Ass Prof, Study Director — Cairo University
Locations (1):
- Faculty of Dentistry, Cairo University, Cairo, Egypt